CLINICAL TRIAL: NCT03721302
Title: A Prospective, Multinational, Observational, Cohort Study Sepsis in Hospitalised Neonates in Areas With High Endemic Levels of Antimicrobial Resistance.
Brief Title: NeoAMR Observational Study in Neonatal Sepsis
Status: Completed | Type: Observational
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: St George's, University of London (Other); PENTA Foundation (Network); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: NeoOBS 001
Record Dates: First submitted 2018-10-04; First posted 2018-10-26 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2018-10

CONDITIONS: Neonatal SEPSIS
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbiological isolates
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main Study Clinical Sepsis: Clinical and Antimicrobial Assessments
  Interventions: Other: Main study clinical sepsis
- Microbiology Sub study: Clinical and Antimicrobial Assessments
  Interventions: Other: Main study clinical sepsis; Other: Microbiology sub study

INTERVENTIONS:
Other: Main study clinical sepsis — No intervention-Observational study
Other: Microbiology sub study — Analysis of Bacterial isolates
  Groups: Microbiology Sub study

SUMMARY:
Prospective, multinational, multicentre, observational cohort study of neonatal sepsis in partner institutions. The cohort study will be designed to evaluate health care utilization and current clinical practice and to assess risk factors for and outcomes of babies with neonatal sepsis (culture-negative and culture-positive).

DETAILED DESCRIPTION:
1. NeoSEPSIS: Consecutive hospitalized babies with neonatal sepsis will be recruited and followed up until discharge from hospital or death (for a maximum of 28 days). A minimal neonatal sepsis dataset will determine (i) clinical presentations, associated features and risk factors (for example prematurity, SGA (small for gestational age)), (ii) rates of culture-positivity among babies with sepsis, (iii) current empirical treatment approaches (antimicrobials selected, dose, etc) (iv) outcomes of sepsis, including death, need for intensive care interventions and recurrence of sepsis during the follow-up period. Microbiological samples will be taken from sterile sites, blood and CSF, as clinically indicated and will be processed locally.
2. NeoBSI: Consecutive babies with positive blood/CSF cultures and sepsis will be recruited. Patient inclusion will be based on identification of relevant specified bacteria from blood / CSF cultures. In addition to the data collected for NeoSEPSIS, information will be collected on the isolates and their antimicrobial susceptibility patterns.

ELIGIBILITY:
Inclusion Criteria:

* In-patient in the hospital (NNU (Neonatal unit) or paediatric ward) of one of the partner institutions

  * Age <60 days of age
  * Clinical suspicion of a new episode of sepsis (as defined below)** together with planned treatment with IV antibiotics OR new episode of confirmed bacterial meningitis^ OR new episode of infection in which a Carbapenem-resistant organism (CRO) is isolated from blood culture OR new episode of infection in which a candida species is isolated from blood culture
  * Informed consent from parent / guardian
  * Willingness to provide location information and to be contacted at 28 days from start of antibiotic treatment

Exclusion Criteria:

* • Previously enrolled in this study, unless readmitted and re-started on antibiotics before the 28 day follow-up limit is reached

  * Enrollment in any interventional trial
  * A serious, non-infective co-morbidity (other than prematurity), anticipated to cause death within 72 hours

Max Age: 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized Babies with significant sepsis
Sampling Method: Non-Probability Sample
Enrollment: 3202 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Mortality Rate | 28 days
  To estimate mortality rates in hospitalised infants less than 60 days of age who are being treated for significant sepsis (where significant is defined as presenting with 2 or more of the signs /symptoms listed in the inclusion criteria).

SECONDARY OUTCOMES:
To determine the microbiological epidemiology, including antimicrobial susceptibility and resistance mechanisms, in infants with positive blood and/or cerebrospinal fluid culture | 28 days
  The incidence of culture positive and culture negative sepsis (both bloodstream and CSF isolates)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Sharland, Principal Investigator — St. George's Hospital, University of London
Locations (19):
- Dhaka Shishu Hospital, Dhaka, Bangladesh
- Brazil (2):
  - FCM da Santa Casa de São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto, São Paulo
- China (3):
  - Beijing Children Hospital, Beijing
  - Beijing Obstetrics and Gynecology Hospital, Beijing
  - Shenzhen Children Hospital, Shenzhen
- Hippokration Hospital, Thessaloniki, Greece
- India (3):
  - King Edward Memorial Hospital and Seth Gordhandas Sunderdas Medical College, Mumbai
  - Lady Hardinge Medical College, New Delhi
  - Jawaharlal Institute of Postgraduate Medical Education and Research (JIPMER), Puducherry
- Bambino Gesu Hospital, Rome, Italy
- KEMRI/Wellcome Trust Research Programme, Kilifi, Kenya
- South Africa (3):
  - Tygerberg Hospital, Cape Town
  - Charlotte Maxeke, Johannesburg
  - Chris Hani Baragwanath Academic Hospital, Johannesburg
- Thailand (2):
  - Queen Sirikit National Institute of Child Health, Bangkok
  - Chiang Rai Prachanukroh Hospital, Chiang Rai
- Mulago Hospital, Kampala, Uganda
- Vietnam National Hospital of Paediatrics, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Folgori L, Ellis SJ, Bielicki JA, Heath PT, Sharland M, Balasegaram M. Tackling antimicrobial resistance in neonatal sepsis. Lancet Glob Health. 2017 Nov;5(11):e1066-e1068. doi: 10.1016/S2214-109X(17)30362-5. No abstract available. PMID 29025624
- [Derived] Russell NJ, Stohr W, Plakkal N, Cook A, Berkley JA, Adhisivam B, Agarwal R, Ahmed NU, Balasegaram M, Ballot D, Bekker A, Berezin EN, Bilardi D, Boonkasidecha S, Carvalheiro CG, Chami N, Chaurasia S, Chiurchiu S, Colas VRF, Cousens S, Cressey TR, de Assis ACD, Dien TM, Ding Y, Dung NT, Dong H, Dramowski A, Ds M, Dudeja A, Feng J, Glupczynski Y, Goel S, Goossens H, Hao DTH, Khan MI, Huertas TM, Islam MS, Jarovsky D, Khavessian N, Khorana M, Kontou A, Kostyanev T, Laoyookhon P, Lochindarat S, Larsson M, Luca M, Malhotra-Kumar S, Mondal N, Mundhra N, Musoke P, Mussi-Pinhata MM, Nanavati R, Nakwa F, Nangia S, Nankunda J, Nardone A, Nyaoke B, Obiero CW, Owor M, Ping W, Preedisripipat K, Qazi S, Qi L, Ramdin T, Riddell A, Romani L, Roysuwan P, Saggers R, Roilides E, Saha SK, Sarafidis K, Tusubira V, Thomas R, Velaphi S, Vilken T, Wang X, Wang Y, Yang Y, Zunjie L, Ellis S, Bielicki JA, Walker AS, Heath PT, Sharland M. Patterns of antibiotic use, pathogens, and prediction of mortality in hospitalized neonates and young infants with sepsis: A global neonatal sepsis observational cohort study (NeoOBS). PLoS Med. 2023 Jun 8;20(6):e1004179. doi: 10.1371/journal.pmed.1004179. eCollection 2023 Jun. PMID 37289666